CLINICAL TRIAL: NCT00048724
Title: PEG-Intron as Maintenance Therapy vs. an Untreated Control Group in Adult Subjects With Compensated Cirrhosis (METAVIR F4), Secondary to Chronic Hepatitis C, Who Have Failed to Respond to Therapy With Any Alpha Interferon Plus Ribavirin
Brief Title: Peg-Intron for Prevention of Disease Progress in Chronic Hepatitis C Patients With Cirrhosis (Study P02569)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02569
Record Dates: First submitted 2002-11-06; First posted 2002-11-08 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Chronic Hepatitis C; Cirrhosis
Keywords: Hepatitis C; Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis; Hepatitis C | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PegIntron (Experimental): PegIntron (peginterferon alfa-2b) 0.5 µg/kg subcutaneously once weekly as maintenance therapy for 60 months with a 4-week post-treatment follow-up
  Interventions: Biological: peginterferon alfa-2b (SCH 54031)
- Untreated Control (No Intervention)

INTERVENTIONS:
Biological: peginterferon alfa-2b (SCH 54031) — 0.5 µg/kg subcutaneously once weekly for 60 months
  Other Names: PegIntron
  Arms: PegIntron

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of PEG-Intron vs. no treatment for the prevention of disease progression in adult subjects with compensated cirrhosis secondary to chronic hepatitis C, who failed to respond to therapy with an a interferon plus ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Age at entry 18-65 years;
* Non-responders to previous treatment (minimum of 3 months) with an alpha interferon plus ribavirin;
* Liver biopsy demonstrating cirrhosis

Exclusion Criteria:

* Any other cause for liver disease other than chronic hepatitis C;
* History or presence of complications of cirrhosis;
* Alcohol or illicit drug abuse or treatment with methadone within the past 2 years;
* Diseases or conditions that could interfere with participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2002-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Bruix J, Poynard T, Colombo M, Schiff E, Burak K, Heathcote EJ, Berg T, Poo JL, Mello CB, Guenther R, Niederau C, Terg R, Bedossa P, Boparai N, Griffel LH, Burroughs M, Brass CA, Albrecht JK; EPIC3 Study Group. Maintenance therapy with peginterferon alfa-2b does not prevent hepatocellular carcinoma in cirrhotic patients with chronic hepatitis C. Gastroenterology. 2011 Jun;140(7):1990-9. doi: 10.1053/j.gastro.2011.03.010. Epub 2011 Mar 17. PMID 21419770

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analysis population is modified intent to treat (MITT), comprising 626 randomized subjects from sites compliant with GCP (Good Clinical Practice). Two sites were closed due to GCP noncompliance, and the 5 subjects from these sites were excluded from analyses.
Groups:
- PegIntron: PegIntron 0.5 µg/kg subcutaneously once weekly as maintenance therapy for 60 months with a 4-week post-treatment follow-up
Period: Overall Study
Arm/Group | PegIntron | Untreated Control
Started | 311 | 315
Completed | 195 | 197
Not Completed | 116 | 118
Not completed — Adverse Event | 53 | 12
Not completed — Withdrawal by Subject | 34 | 54
Not completed — Lost to Follow-up | 5 | 5
Not completed — Protocol-defined Clinical Event | 17 | 32
Not completed — Noncompliance With Protocol | 4 | 12
Not completed — Did Not Meet Protocol Eligibility | 2 | 2
Not completed — Administrative | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PegIntron | Untreated Control | Total
Number analyzed (Participants) | 311 | 315 | 626
Age, Customized [Number; unit: Participants]
  <=50 years | 130 | 132 | 262
  >50 years | 181 | 183 | 364
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 100 | 205
  Male | 206 | 215 | 421

OUTCOME MEASURES:

1. Primary Outcome: Time to Observation of the First Clinical Event Experienced by a Subject
Description: Clinical events are liver decompensation [variceal bleeding, development of Child-Pugh Class C, hepatic encephalopathy ≥Grade 2, ascites], hepatic carcinoma, death, and/or liver transplantation
Time Frame: Up to 60 months of treatment or observation, or when 98 subjects experience at least one clinical event
Population: Analysis population is modified intent to treat (MITT), comprising all randomized subjects from sites compliant with GCP (Good Clinical Practice). Two sites were closed due to GCP noncompliance, and the 5 subjects from these sites were excluded from efficacy analyses.
Measure: Number; unit: Participants
Arm/Group | PegIntron | Untreated Control
Number analyzed (Participants) | 311 | 315
Participants
  <=6 Months | 3 | 2
  >6 to 12 Months | 5 | 5
  >12 to 18 Months | 4 | 4
  >18 to 24 Months | 3 | 7
  >24 to 30 Months | 7 | 6
  >30 to 36 Months | 1 | 6
  >36 to 42 Months | 0 | 5
  >42 to 48 Months | 2 | 0
  >48 to 54 Months | 2 | 1
  >54 to 60 Months | 0 | 0
  Total Over Study | 27 | 36
Statistical Analysis 1: Comparison: PegIntron vs Untreated Control; The primary scientific hypothesis is that, 0.5 ug/kg subcutaneous once weekly PegIntron as maintenance therapy is efficacious, when compared to no treatment, in the prevention of clinical events in adult subjects with compensated cirrhosis (Metavir F4), secondary to Chronic Hepatitis C, who have failed to respond to therapy with any α interferon plus ribavirin; Test type: Superiority or Other; p = 0.1439, Cox Proportional Hazards Model; Age (<= 50 years, >50 years) and participation in a prior study (yes, no) were stratification factors; Hazard Ratio (HR) = 1.452, 95% CI [0.880 to 2.396] — Hazard ratio represents results of untreated control relative to treatment

2. Secondary Outcome: Time to Observation of the Disease Progression Experienced by a Subject
Description: Disease progression was observation of any clinical event defined for the primary outcome, plus any of development of Child-Pugh Class B, emergence of varices, or enlargement of pre-existing varices requiring additional therapy.
Time Frame: Up to 60 months of treatment or observation, or when 98 subjects experience at least one clinical event
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | PegIntron | Untreated Control
Number analyzed (Participants) | 311 | 315
Participants
  <=6 Months | 16 | 17
  >6 to 12 Months | 6 | 6
  >12 to 18 Months | 5 | 7
  >18 to 24 Months | 12 | 20
  >24 to 30 Months | 10 | 11
  >30 to 36 Months | 4 | 9
  >36 to 42 Months | 2 | 4
  >42 to 48 Months | 2 | 6
  >48 to 54 Months | 5 | 4
  >54 to 60 Months | 1 | 3
  Total Over Study | 63 | 87
Statistical Analysis 1: Comparison: PegIntron vs Untreated Control; The secondary hypothesis is that 0.5 ug/kg subcutaneous once weekly PegIntron as maintenance therapy is efficacious, when compared to no treatment, in the prevention of disease progression in adult subjects with compensated cirrhosis (Metavir F4), secondary to Chronic Hepatitis C, who have failed to respond to therapy with any α interferon plus ribavirin; Test type: Superiority or Other; p = 0.0070, Cox Proportional Hazards Model; Age (<= 50 years, >50 years) and participation in a prior study (yes, no) were stratification factors; Hazard Ratio (HR) = 1.564, 95% CI [1.130 to 2.166] — Hazard ratio represents results of untreated control relative to treatment

ADVERSE EVENTS:
Arm/Group | PegIntron | Untreated Control
Serious Adverse Events (participants affected / at risk) | 93/311 | 74/315
Other Adverse Events (participants affected / at risk) | 290/311 | 260/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron (N=311) | Untreated Control (N=315)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5) | 1 (2)
AUTOIMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 1 (1)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
CATARACT NUCLEAR (Eye disorders) | 1 (1) | 0 (0)
DIABETIC RETINOPATHY (Eye disorders) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0)
VITREOUS HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 3 (3)
ASCITES (Gastrointestinal disorders) | 1 (1) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 1 (2)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HERNIAL EVENTRATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 10 (10)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1)
PERITONITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL FISSURE (Gastrointestinal disorders) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 0 (0) | 4 (8)
CHEST PAIN (General disorders) | 2 (2) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (3) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 1 (1)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 3 (3) | 3 (3)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 4 (4) | 0 (0)
CHRONIC HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 2 (2)
HEPATIC MASS (Hepatobiliary disorders) | 1 (1) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 2 (2) | 0 (0)
PORTAL HYPERTENSIVE GASTROPATHY (Hepatobiliary disorders) | 0 (0) | 1 (1)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 2 (2) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
BRONCHIECTASIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 4 (4) | 0 (0)
HAEMOPHILUS SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
MENINGITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
PILONIDAL CYST (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 4 (4) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PSOAS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 2 (3) | 0 (0)
RECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
NECK INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL FISTULA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND SECRETION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALPHA 1 FOETOPROTEIN INCREASED (Investigations) | 0 (0) | 3 (3)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
TRANSPLANT EVALUATION (Investigations) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
DIABETES WITH HYPEROSMOLARITY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
EXTRASKELETAL OSSIFICATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 12 (12)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT PALATE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SALIVARY GLAND ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL CYST (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 2 (2)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 2 (2) | 2 (2)
HYPERTONIA (Nervous system disorders) | 1 (1) | 0 (0)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 1 (1)
MENINGORRHAGIA (Nervous system disorders) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (3) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 3 (3) | 1 (1)
BRADYPHRENIA (Psychiatric disorders) | 0 (0) | 1 (1)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
CALCULUS URINARY (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (2) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BREAST CALCIFICATIONS (Reproductive system and breast disorders) | 2 (2) | 0 (0)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 2 (2) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
MIDDLE LOBE SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
POST PROCEDURAL DRAINAGE (Surgical and medical procedures) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) | 0 (0)
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 0 (0) | 2 (2)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2) | 1 (1)
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 (0) | 1 (1)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 0 (0)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 (0) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 1 (1)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron (N=311) | Untreated Control (N=315)
LEUKOPENIA (Blood and lymphatic system disorders) | 20 (31) | 8 (9)
NEUTROPENIA (Blood and lymphatic system disorders) | 43 (119) | 18 (26)
SPLENOMEGALY (Blood and lymphatic system disorders) | 60 (69) | 54 (61)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 52 (122) | 20 (41)
ABDOMINAL PAIN (Gastrointestinal disorders) | 33 (40) | 21 (27)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 45 (66) | 46 (67)
CONSTIPATION (Gastrointestinal disorders) | 16 (20) | 14 (17)
DIARRHOEA (Gastrointestinal disorders) | 37 (57) | 25 (30)
DYSPEPSIA (Gastrointestinal disorders) | 20 (27) | 21 (29)
GASTRITIS (Gastrointestinal disorders) | 20 (22) | 40 (42)
NAUSEA (Gastrointestinal disorders) | 49 (62) | 39 (58)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 35 (41) | 52 (56)
VOMITING (Gastrointestinal disorders) | 18 (21) | 11 (11)
ASTHENIA (General disorders) | 45 (70) | 37 (48)
CHILLS (General disorders) | 26 (37) | 3 (4)
FATIGUE (General disorders) | 103 (152) | 78 (92)
INFLUENZA LIKE ILLNESS (General disorders) | 46 (61) | 4 (4)
INJECTION SITE ERYTHEMA (General disorders) | 36 (37) | 0 (0)
IRRITABILITY (General disorders) | 41 (48) | 17 (18)
MALAISE (General disorders) | 16 (41) | 11 (13)
OEDEMA PERIPHERAL (General disorders) | 19 (23) | 29 (39)
PYREXIA (General disorders) | 57 (163) | 14 (15)
HEPATOMEGALY (Hepatobiliary disorders) | 45 (61) | 51 (62)
BRONCHITIS (Infections and infestations) | 20 (28) | 23 (38)
INFLUENZA (Infections and infestations) | 16 (18) | 28 (37)
NASOPHARYNGITIS (Infections and infestations) | 20 (27) | 25 (36)
SINUSITIS (Infections and infestations) | 17 (23) | 17 (20)
URINARY TRACT INFECTION (Infections and infestations) | 9 (20) | 16 (22)
ANOREXIA (Metabolism and nutrition disorders) | 25 (32) | 8 (10)
DECREASED APPETITE (Metabolism and nutrition disorders) | 21 (27) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 68 (120) | 63 (90)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 44 (47) | 39 (51)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 29 (38) | 17 (19)
MYALGIA (Musculoskeletal and connective tissue disorders) | 76 (242) | 19 (22)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 23 (36) | 13 (14)
DIZZINESS (Nervous system disorders) | 22 (32) | 20 (23)
HEADACHE (Nervous system disorders) | 103 (249) | 47 (62)
ANXIETY (Psychiatric disorders) | 24 (46) | 16 (19)
DEPRESSION (Psychiatric disorders) | 35 (41) | 26 (35)
INSOMNIA (Psychiatric disorders) | 50 (77) | 45 (55)
RENAL CYST (Renal and urinary disorders) | 6 (7) | 19 (19)
COUGH (Respiratory, thoracic and mediastinal disorders) | 33 (46) | 34 (46)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 14 (15)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 23 (30) | 9 (9)
ALOPECIA (Skin and subcutaneous tissue disorders) | 36 (41) | 27 (30)
PRURITUS (Skin and subcutaneous tissue disorders) | 42 (64) | 27 (38)
RASH (Skin and subcutaneous tissue disorders) | 31 (41) | 10 (14)
SPIDER NAEVUS (Skin and subcutaneous tissue disorders) | 14 (16) | 17 (19)
HYPERTENSION (Vascular disorders) | 41 (47) | 38 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide review copies to the sponsor 30 days prior to submission for publication or presentation. The sponsor shall have editorial rights and the right to review and comment on the data analysis and presentation. If the parties disagree, investigator agrees to meet with the sponsor's representatives for the purpose of making good faith efforts to discuss and resolve any such issues.